CLINICAL TRIAL: NCT02589535
Title: Circulating Stem Cells, SDF-1, HIF-1 and Sepsis: Relationship Between Indices of Sepsis and Emergency Abdominal Surgical Patients
Brief Title: Circulating Stem Cells, SDF-1, HIF-1 and Sepsis's Indices in Emergency Abdominal Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Foggia (Other)
Collaborators: Fondo di Sviluppo e Coesione 2007-2013 APQ RicercaRegionePuglia FutureInResearch (Unknown)
Responsible Party: Principal Investigator, Cotoia Antonella, Aggregate Professor, PhD, University of Foggia
Other Study IDs: 69/CE/2015
Record Dates: First submitted 2015-10-24; First posted 2015-10-28 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- septic: Group Gb: postoperative septic patients in intensive care unit (ICU)] Gb1: the group of septic patients treated with extracorporeal hemoperfusion therapy and conventional therapy according to the Surviving Sepsis Campaign guidelines Gb2 group treated with conventional therapy according to the Surviving Sepsis Campaign guidelines
- no septic: Ga: postoperative patients in emergency surgical ward (ES)
- healthy: Healthy people

SUMMARY:
Septic shock is a systemic inflammatory response syndrome with acute circulatory failure secondary to a documented infection. It is the most feared complication in ICU patients, with a 50% mortality rate.

The study of stem cells and their experimental use in sepsis treatment is particularly relevant in the international scientific research, where Italy plays an important role. In the vast and complex field of stem cell research, the primary aim of the current proposal is to evaluate the time course level of circulating endothelial progenitor stem cells CD34 + / CD133 + (EPCs), and some factors EPCs-related, such as hypoxia- inducible factor (HIF- 1) and stromal derived factor-1 (SDF-1) in septic patients undergoing major abdominal surgery.

Secondary objective 2: to investigate the relationship between CD133/CD34, HIF-1, SDF-1a and outcome of septic/septic shock patients treated with standard conventional therapy alone (CT) or with extracorporeal hemoperfusion therapy (HCT).

DETAILED DESCRIPTION:
Primary objective: to determine the time course level of the circulating EPC (CD133/CD34), SDF-1a, and HIF-1 in septic patients undergoing major abdominal surgery.

Secondary objective 1: to investigate the relationship between these factors: CD133/CD34, HIF-1 and SDF-1a.

Secondary objective 2: to investigate the relationship between CD133/CD34, HIF-1, SDF-1° and outcomeof septic/septic shock patients treated with standard conventional therapy alone (CT) or with extracorporeal hemoperfusion therapy (HCT).

In this trial, we hypothesize that CD133/CD34, HIF1 and SDF1a will increase in septic surgical patients as consequence of impaired tissue perfusion and cellular hypoxia. Our hypothesis is based on the fact that the stimulation of factors hypoxia-related, as SDF-1a and HIF-1 could be the primary step for bone marrow stem cells stimulation. Furthermore, we assume that survivors septic patients will show higher levels of EPC, HIF-1 and SDF-1a.

Each day, the anesthesiologist of the operating room and the on-call anesthesiologist will alerts the principal investigator to a potential eligible patient. Participants included in the trial will be divided into two groups:

* C group: postoperative non septic patients in emergency surgical ward (ES) (control group)
* S group: postoperative septic shock patients in intensive care unit (ICU) Healthy volunteers (H group) will be recruited from among staff members of the University Hospital of Foggia

The research study can provide useful parameters for early diagnostic and therapeutic interventions in sepsis which is the leading cause of death from infection, with an incidence of approximately 10% in ICU postoperative patients according to recent epidemiologic studies.

ELIGIBILITY:
Inclusion criteria:

Caucasian, Over 18 years of age

Exclusion criteria:

when it is impossible to collect blood samples (organizational reasons or because of emergencies regarding the health of the patients),Pregnant patients,Organ transplantation, Palliative care,Metastatic cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: postoperative patients undergoing major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
time course level of circulating endothelial progenitor stem cells CD133+/CD34+, HIF1 and SDF in septic patients undergoing emergency major abdominal surgery. | 1-10 days after intervention
  to determine the time course level of the circulating EPC (CD133/CD34), SDF-1a, and HIF-1 in septic patients undergoing major abdominal surgery.

SECONDARY OUTCOMES:
correlation among time course level of circulating stem cells, hypoxia-inducible factor-1 (HIF-1) and stromal derived factor - 1 (SDF-1) | 1-10 days after intervention
  to investigate the relationship between these factors: CD133/CD34, HIF-1 and SDF-1a.
relationship between CD133/CD34, HIF-1, SDF-1a and outcome. | 1-10 days after intervention
  to investigate the relationship between CD133/CD34, HIF-1, SDF-1a and outcome of patients treated with conventional therapy alone or plus extracorporeal hemoperfusion therapy

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Cotoia, MD, PhD, Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- University of Foggia, Foggia, Italy

REFERENCES:
- [Result] Friedrich EB, Walenta K, Scharlau J, Nickenig G, Werner N. CD34-/CD133+/VEGFR-2+ endothelial progenitor cell subpopulation with potent vasoregenerative capacities. Circ Res. 2006 Feb 17;98(3):e20-5. doi: 10.1161/01.RES.0000205765.28940.93. Epub 2006 Jan 26. PMID 16439688
- [Result] Cribbs SK, Martin GS, Rojas M. Monitoring of endothelial dysfunction in critically ill patients: the role of endothelial progenitor cells. Curr Opin Crit Care. 2008 Jun;14(3):354-60. doi: 10.1097/MCC.0b013e3282fc216d. PMID 18467899
- [Result] Kalil AC, Florescu MC. Blood purification: can we purify our patients from sepsis? Crit Care Med. 2013 Sep;41(9):2244-5. doi: 10.1097/CCM.0b013e318291cad5. No abstract available. PMID 23979379
- [Derived] Cotoia A, Cela O, Palumbo G, Altamura S, Marchese F, Mangialetto N, La Bella D, Lizzi V, Capitanio N, Cinnella G. High mobilization of CD133+/CD34+ cells expressing HIF-1alpha and SDF-1alpha in septic abdominal surgical patients. BMC Anesthesiol. 2020 Jun 27;20(1):158. doi: 10.1186/s12871-020-01068-w. PMID 32593288
- [Derived] Cotoia A, Mirabella L, Altamura S, Villani R, Marchese F, Ferrara G, Mariano K, Livio T, Cinnella G. Circulating stem cells, HIF-1, and SDF-1 in septic abdominal surgical patients: randomized controlled study protocol. Trials. 2018 Mar 12;19(1):179. doi: 10.1186/s13063-018-2556-0. PMID 29530072